CLINICAL TRIAL: NCT02349035
Title: Application of Targeted Reinnervation for People With Transradial Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); San Antonio Military Medical Center (U.S. Federal Agency); Northwestern University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Todd Kuiken, Director, Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00101444; R01HD081525-01 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-28 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Amputation; Traumatic, Hand, and Wrist; Amputation; Traumatic, Hand, at Wrist Level
Keywords: Transradial amputee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMR surgery to evaluate pattern recognition control (Experimental): Perform Targeted Muscle Reinnervation (TMR) surgery and evaluate transradial TMR pattern recognition control of multifunctional prostheses.
  Interventions: Device: Compare control of multifunction transradial prosthesis; Procedure: Perform TMR surgery and evaluate transradial TMR pattern recognition control of multifunctional prostheses.

INTERVENTIONS:
Device: Compare control of multifunction transradial prosthesis — Subjects practice control methods using a VR system. EMG data and virtual games are used and provide data to assess control methods without prosthesis. Subjects are fit with commercially available multifunctional hand system. They receive 1-3 days of training for conventional or pattern recognition control. They return home for an 8 week trial. They use the prosthesis for 2 hours a day across the 8 week trial. They keep a log of use and check with a therapist about usage and performance. After the 8 week trial, data from the prosthesis is downloaded. The subject will complete 1-3 days of outcomes testing. They perform a series of tests and data is recorded. The subject will repeat the 1-3 days of training, 8 week home trial, and 1-3 days of outcomes testing with either type of control.
Procedure: Perform TMR surgery and evaluate transradial TMR pattern recognition control of multifunctional prostheses. — Subject has Targeted Muscle Reinnervation surgery. The surgery transfers median nerve to flexor digitorum superficialis muscle and ulnar nerve to flexor carpi ulnaris muscle. Two weeks after surgery, exercises start for muscle recovery. Then return to prosthesis from Phase 1 for 6 months. If they have pattern recognition control, usage and performance will be tracked for 6 months. If they return to conventional control, they will not complete tests, track usage, or performance. Six months after surgery, they return to pattern recognition control. Receive 1-3 days of training. Take prosthesis home for 8 week trial. Log use of device, note issues, and follow up with therapist. After home trial, 1-3 days of outcomes testing are completed and usage data downloaded. Continue using their prostheses for an additional 3-4 months. At 12 months after surgery, a final round of 1-3 days of testing and data are downloaded.

SUMMARY:
The purpose of this study is to improve prosthesis control for transradial amputees with combining targeted muscle reinnervation surgery (TMR) and pattern recognition control.

DETAILED DESCRIPTION:
Phase 1: Transradial amputees will be asked to come to the Rehabilitation Institute of Chicago, Walter Reed National Military Medical Center or the San Antonio Military Medical Center for initial fitting with a prosthetist for a multifunctional hand system or multifunctional hand and wrist system. The prosthesis system will consist of a custom-made socket and commercially available components. The first visit (up to five days)s involves casting, creating and fitting of a socket that will be used for the study. During the initial and subsequent visits, the subject will be asked asked to practice various control methods using a virtual reality system. EMG data and virtual "games" will be used to practice the control and will provide quantitative data that can be used to assess the various control methods mathematically, without the prosthesis.

Once they receive a socket, they will complete 1-3 days of training to learn how to control the prosthesis with either conventional or pattern recognition control. The prosthetic training days may occur concurrently with the fitting appointment or it may require a separate visit. The subject will return home for the initial 8 week home use trial. They will be asked to use the prosthesis for an average of 2 hours per day across the 8 week home trial period. They will keep a home log of prosthesis use and check in weekly with a therapist to discuss usage and prosthesis performance. They may also be provided with a laptop computer with a camera for Skyping. The laptop can be connected to the prosthesis, and the screen can be viewed remotely. The research team can then continue with remote follow up with more training and problem solving as needed. Directly following the 8 week home trial period, usage data from the prosthesis will be downloaded. The subject will complete 1-3 days of outcomes testing with a therapist. A series of tests will be performed and data recorded of your performance. The subject will then repeat the 1-3 days of training, 8 week home trial period, and 1-3 days of outcomes testing with either the other type of control (i.e. conventional or pattern recognition).

Phase 2: The subject will return to one of the three centers for Targeted Muscle Reinnervation (TMR) surgery. The surgery is an outpatient procedure that will be performed under general anesthesia, consistent with current standard of care. The surgery will involve the transfer of the median nerve to the flexor digitorum superficialis (DFS) muscle and the ulnar nerve will be transferred to the flexor carpi ulnaris (FCU) muscle. Both transfers can be done with a single incision. Alternative target muscles (e.g. the brachioradialis muscle) can be used if trauma interferes with use of the DFS and/or FCU. Some post-operative pain is expected and the subject will be given a prescription for pain medication if needed. Two weeks after the surgery the subject will be asked to start doing exercises to help with muscle recovery. They will return to using the prosthesis from Phase 1 with either conventional or pattern recognition control for 6 months after surgery. Socket adjustments will be made if needed. If they return to using pattern recognition control, their usage and performance data will be tracked during this 6 month period. The subject may be provided with a laptop computer and asked to perform a series of virtual tests. They will receive additional training on how to complete these tests. If the subject returns to using conventional control, they will not be asked to complete the additional tests, nor will the usage or performance data be tracked. Six months after surgery, when reinnervation of the target muscles has been completed, the subject will return to using the prosthesis with pattern recognition control. They will be asked to return to one of the three centers if socket adjustments or a replacement socket is needed. The subject will receive 1-3 days of pattern recognition control training, only this time special attention will be paid to utilizing EMG from target muscles for improved function. Preliminary testing will be done to ensure that they can adequately use the prosthesis. The subject will then take the prosthesis home for a third 8-week home-use trial. The subject will be asked to log daily use of the device, note any issues, and follow up weekly with a therapist. After this home-use trial, the same 1-3 days of comprehensive outcomes testing will be completed and usage data from their prostheses will be downloaded.

Finally, the subject will continue using the prostheses at home for an additional 3-4 months. No usage requirements will be given during this time. At the end of this 3-4 month period (approximately 12 months after surgery), they will have a final round of 1-3 days of testing with the complete toolbox and data from the prosthesis will be downloaded.

The days of prosthesis training and testing may take place at the Rehabilitation Institute of Chicago, Walter Reed National Military Medical Center, or the San Antonio Military Medical Center or near your home. Study coordinators will determine the best location.

ELIGIBILITY:
Inclusion Criteria:

* A upper limb amputation at the transradial level

Exclusion Criteria:

* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant user feedback through questionnaires and informal discussion adds significant value to this study.
* Significant other co morbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2020-12 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Improve pattern recognition control of multifunction prostheses for transradial amputees. | 15 months from initial enrollment
  Improved control of prosthesis as seen through functional use improvements.

SECONDARY OUTCOMES:
Modified Box and Blocks | At 2 and 4 months pre-op; At 6 and 10 months post-op
  Timed task to assess prosthetic control.
Clothespin Relocation Test | At 2 and 4 months pre-op; At 6 and 10 months post-op
  Timed task to assess prosthetic control.
ACMC | At 2 and 4 months pre-op; At 6 and 10 months post-op
  Assessment of capacity for myoelectric prosthetic control
Jebsen Test of Hand Function | At 2 and 4 months pre-op; At 6 and 10 months post-op
  7 part timed diagnostic test to determine the level of hand function.
Southampton Hand Assessment Procedure (SHAP) | At 2 and 4 months pre-op; At 6 and 10 months post-op
  The test consists of the manipulation of a series of both lightweight and heavyweight abstract objects. The procedure is designed to provide a score of functionality.
OPUS-UEFS | At 2 and 4 months pre-op; At 6 and 10 months post-op
  An instrument that evaluates the activity limitations, quality of life, and patient satisfaction with services and devices.
Activities Measure for Upper Limb Amputees (AM-ULA) | At 2 and 4 months pre-op; At 6 and 10 months post-op
  A clinician rated measure of an upper limb amputee's performance of daily functional activities using a prosthesis.
TAC TEST/ Motion Test | At 2 and 4 months pre-op; At 6 and 10 months post-op
  Virtual reality testing of classification accuracy, motion completion rate, motion completion time and path efficiency.
PSFS | At 2 and 4 months pre-op; At 6 and 10 months post-op
  Used to assess functional ability to complete specific activities

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Kuiken, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (3):
- United States (3):
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - San Antonio Military Medical Center, Fort Sam Houston, Texas